CLINICAL TRIAL: NCT04618991
Title: Assessment of the Impact on the Quality of Life of Surgically Assisted Maxillary Expansion in Adult Patients Followed for Obstructive Sleep Apnea Syndrome
Acronym: QUAVIMAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP201080
Record Dates: First submitted 2020-10-15; First posted 2020-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; quality of life; surgically assisted rapid maxillary expansion; distraction osteogenesis; palatal expansion technique
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with SAHOS for whom maxillary transversal surgery (Experimental): Adult patients with SAHOS for whom maxillary transversal surgery is recommended.
  Interventions: Other: Filling the Quebec Sleep Questionnaire

INTERVENTIONS:
Other: Filling the Quebec Sleep Questionnaire — Filling the Quebec Sleep Questionnaire (QSQ) by the pre-surgery patient, then at 3 months post surgery and 1 year post surgery.

SUMMARY:
The research aims to assess the impact on quality of life of surgically maxillary expansion in adult patients followed for obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
This assessment will be done using the following elements:

* The score of the Quebec sleep questionnaire (QSQ), developed in 2004 by Lacasse Y. et al. This questionnaire is specific to sleep apnea and may be self-administered. The main interest of this questionnaire is to measure the change in quality of life over time.
* The Epworth Scale Score, developed in 1991 by Murray W. John. This is a self-administered questionnaire developed to measure daytime sleepiness.
* Gender, age group, BMI
* The radiological assessment
* The results of polysomnography

Patients will be followed for a period of 1 year and one month after surgery. The protocol visits correspond to the rhythm of post-surgery follow-up consultations in current practice.

These patients are followed by Dr. Pételle at Saint-Antoine Hospital. During these visits, they will complete the Quebec sleep questionnaire and the Epworth scale, at baseline, at 3 months and then at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* With obstructive sleep apnea confirmed by polysomnography
* Surgical indication for surgically maxillary expansion

Exclusion Criteria:

* - Patients refusing to participate in the survey having formulated their opposition
* Diabetes,
* Obesity (BMI> 30)
* Failure to provide informed written consent
* Refusal or inability to return to all follow-up visits and sleep studies
* Patient pregnant or planning to become pregnant in the next 12 months or breastfeeding
* Surgical resection or radiation therapy for cancer or congenital malformations of the larynx, tongue or throat (Note that some previous surgeries, such as uvulopalatopharyngoplasty (UPPP), tonsillectomy or adenoidectomy, to remove obstructions related to obstructive sleep apnea are allowed)
* Obvious obstructions of the fixed upper airways (tumors, polyps or nasal obstruction)
* Patients who have undergone previous surgery on the mandible and / or maxilla, other than dental treatment.
* Patients included in another clinical study (excluding registers).
* Patients taking medicines such as opiates which may affect sleep, alertness or breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Score of the QSQ | at 3 months
  Score of the QSQ filled directly by the patient before surgery, compared to that then 3 months after surgery.

SECONDARY OUTCOMES:
Score of the Quebec Sleep Questionnaire (QSQ) | at 1 year
  Score of the QSQ filled directly by the patient before surgery, compared to that then 1 year after surgery.
Polysomnography | at 3 months
  Search for a modification of the polysomnography data before and after surgery
Epworth scale | at 1 year
  Epworth scale score changes before and after surgery
correlation between the results of the Quebec Sleep Questionnaire (QSQ) score and the anthropometric data | at 1 year
  correlation between the results of the QSQ score and the anthropometric data

CONTACTS AND LOCATIONS:
Overall Officials: Boris Petelle, Study Chair — Assistance Publique - Hôpitux de Paris
Locations (1):
- Service d'ORL, Hôpital Saint Antoine, Paris, France